CLINICAL TRIAL: NCT00247104
Title: The Use of Cranberries in Women With Preterm Premature Rupture of Membranes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CRANBERRIES-HMO-CTIL
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2006-03

CONDITIONS: Fetal Membranes, Premature Rupture; Premature Birth
Keywords: Urinary tract infection; Endometritis; Respiratory Distress Syndrome; Necrotizing enterocolitis; Intraventricular hemorrhage; Latent period; Neonatal infection
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Premature Birth; Urinary Tract Infections; Endometritis; Respiratory Distress Syndrome; Enterocolitis, Necrotizing

INTERVENTIONS:
Drug: Cranberries - Vaccinium macrocarpon

SUMMARY:
Cranberries have been proved to reduce the rate of urinary tract infections in a population of women with recurrent urinary tract infections in previous studies. The purpose of the study is to examine the efficacy of cranberries in pregnant women with preterm premature rupture of membranes in a)prolonging the latent period (=the time period between the time the water broke and delivery of the fetus) and b)reduction of infectious morbidity of both the mother and infant.

DETAILED DESCRIPTION:
Preterm premature rupture of membranes (PPROM) complicates 2-3.5% of pregnancies and precipitates labor in 30-40% of preterm deliveries. The common practice in early PPROM with no evidence of chorioamnionitis is admission for close surveillance, antibiotic treatment and steroids for fetal lung maturation (until 32 weeks gestation. Intraamniotic infection is evident in up to 75% of women who develop labor during admission. The infection is for the most an ascending infection.

Cranberries have been recognized by the American Indians as a natural means for preventing urinary tract infection. The mechanism of action includes acidification of urine and inhibition of adhesion of pili-harboring bacteria to the transitional epithelium of the urinary tract.

We assume that cranberries will lower the rate of maternal urinary tract infection. Moreover, the active ingredients will pass transplacentally to the fetus, will be secreted in its urine hence, in the amniotic fluid. The active substances would coat the vagina and bring about their effect also in that environment. Having in mind that most if not all chorioamnionitis infections are caused by ascending infection, the cranberries might lengthen the latent period and reduce infectious maternal and neonatal morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Proven premature rupture of membranes
* less than 35 weeks of gestation with good obstetrical dating
* no suspicion of amnionitis
* signed informed consent

Exclusion Criteria:

* Known sensitivity / allergy to cranberries
* Women treated with warfarin
* Drug intolerance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-05; Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
Length (in days) of the latent period
Neonatal infection
Respiratory distress
Admission to NICU (in days)
Neonatal complications rate (NEC, IVH etc)
Maternal infections (uterus, UTI)

SECONDARY OUTCOMES:
Urinary and vaginal flora before and after treatment
Vaginal pH before and after treatment
Amniotic fluid pH before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Drorit Hochner-Celnikier, MD, Study Director — Hadassah Medical Organization; Uriel Elchalal, MD, Study Director — Hadassah Medical Organization; Hagit Daum, MD, Principal Investigator — Hadassah Medical Organization; Shay Porat, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Jepson RG, Mihaljevic L, Craig J. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2004;(2):CD001321. doi: 10.1002/14651858.CD001321.pub3. PMID 15106157
- [Derived] Williams G, Stothart CI, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Nov 10;11(11):CD001321. doi: 10.1002/14651858.CD001321.pub7. PMID 37947276
- [Derived] Williams G, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Apr 17;4(4):CD001321. doi: 10.1002/14651858.CD001321.pub6. PMID 37068952